CLINICAL TRIAL: NCT04144114
Title: The Effect of ProHydrolase® on the Amino Acid, Intramuscular Anabolic Signaling, and Endocrine Response to Resistance Exercise in Trained Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deerland Enzymes (Industry)
Collaborators: Lipscomb University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro18
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Amino Acids
Keywords: Amino Acids; Intramuscular Anabolic Signaling; Endocrine Response; Resistance Training
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey + ProHydrolase® (Experimental): Subjects received 250mg of ProHydrolase® along with 25g of whey protein mixed in a drink every visit for 4 weeks
  Interventions: Dietary Supplement: ProHydrolase®
- Whey (Active Comparator): Subjects received 25g whey protein in a drink every visit for 4 weeks
  Interventions: Dietary Supplement: Whey protein
- Placebo (Placebo Comparator): Subjects received 25g maltodextrin in a drink every visit for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ProHydrolase® — Subjects received 250mg of ProHydrolase® with 25g whey protein mixed together in a drink
  Arms: Whey + ProHydrolase®
Dietary Supplement: Whey protein — Subjects received 25g of whey protein powder mixed to together in a drink
  Arms: Whey
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To examine the amino acid absorption following acute resistance exercise between three supplemental treatments: 1) Whey Protein + ProHydrolase (WPH) 2) Whey Protein (W) and 3) Non-Caloric Placebo (PL). To examine three supplemental treatments (WPH, W, PL) in conjunction with acute resistance exercise on the mTORC1 complex pathway. To examine three supplemental treatments (WPH, W, PL) in conjunction with acute resistance exercise on circulating concentrations of endocrine biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* • At least one-year of resistance training experience

  * Free of any physical limitations (determined by health and activity questionnaire).
  * Between the ages of 18 and 35.
  * Ability to leg press a weight equivalent to 1.5 times their body mass

Exclusion Criteria:

* • Inability to perform physical exercise (determined by health and activity questionnaire)

  * Taking any other nutritional supplement or performance enhancing drug (determined from health and activity questionnaire).
  * Physical injury preventing the athlete from participating in offseason training
  * Any chronic illness that causes continuous medical care

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Amino acid absorption | 4 weeks
  To examine the amino acid absorption following acute resistance exercise between three supplemental treatments: 1) Whey Protein + ProHydrolase (WPH) 2) Whey Protein (W) and 3) Non-Caloric Placebo (PL)
mTORC1 pathway | 4 weeks
  To examine three supplemental treatments (WPH, W, PL) in conjunction with acute resistance exercise on the mTORC1 complex pathway
Endocrine markers | 4 weeks
  To examine three supplemental treatments (WPH, W, PL) in conjunction with acute resistance exercise on circulating concentrations of endocrine biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Lipscomb University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No